CLINICAL TRIAL: NCT05796297
Title: Clinical Impact of Patient Ventilator Asynchrony in Patients With Chronic Respiratory Failure on Long-term Ventilation : a Prospective, Monocentric, Open-label Epidemiological Study
Brief Title: Clinical Impact of Patient-ventilator Asynchrony
Acronym: INSPIRER
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0099
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Chronic Respiratory Failure; Non-invasive Ventilation; Asynchrony Between Patient and Ventilator; Efficacy and Tolerance of Non-invasive Ventilation; Clinical Repercussions of the Various Patient-ventilator Asynchronies
Keywords: Tolerance; Efficiency; Patient ventilator asynchrony; NIV
MeSH Terms: conditions — Patient-Ventilator Asynchrony

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with significant patient ventilator asynchrony: Active Comparator
  Interventions: Device: Transcutaneous Capnography
- Patient without significant patient ventilator asynchrony: Active Comparator
  Interventions: Device: Transcutaneous Capnography

INTERVENTIONS:
Device: Transcutaneous Capnography — Transcutaneous Capnography will be realized at patient home to monitoring nocturnal concentration of carbon dioxide during nocturnal sleeping ventilation

SUMMARY:
The investigator wish to carry out this study to explore the link between patient-ventilator asynchrony with the efficiency and tolerance of NIV but also the quality of life in patients with chronic respiratory failure on long-term ventilation.

DETAILED DESCRIPTION:
Chronic respiratory failure (CRF) is an advanced stage of many respiratory diseases marked by an inability of the respiratory system to ensure vital gas exchange. It affects approximately 3.6 million people in France.

Non-invasive ventilation (NIV) remains the reference treatment in hypercapnic respiratory failure because it reduces inspiratory muscles's work and promotes alveolar ventilation.

The establishment of the NIV is carried out most of the time following an episode of acute decompensation revealing an underlying CRF. It is carried out and supervised in hospital departments to optimize the understanding and adherence of the patient to his illness and his treatment.

Thus, monitoring is a key to measure the tolerance and effectiveness of ventilation. Classically, it is based on multi-year medical consultations, blood gases and nocturnal oximetry. In recent years, the reading of detailed data from software integrated into NIV machines has been increasingly used in current practice in association with the monitoring tools already recommended. It provides additional detailed information on compliance, leaks, apnea-hypopnea index (AHI), obstructive events and asynchrony between the patient and their ventilator.

Many patient-ventilator asynchronies have been described in studies with a negative impact on the quality of ventilation, the quality of sleep under NIV and an increased risk of mortality. However, not all asynchronies have the same consequences and are not all felt by the patient

ELIGIBILITY:
Inclusion Criteria :

* Women and Men aged of at least 18 years old.
* NIV equipment since 6 months ( at least)
* Chronic respiratory failure requiring NIV equipment defined by clinical symptoms (asthenia, excessive daytime sleepiness, headache, dyspnea) and:

In case of obstructive diseases :

Daytime hypercapnia (PaCO2 > 55 mmHg) or Daytime hypercapnia between 50-54 mmHg associated with nocturnal desaturations (at least 5 min below 88% saturation) or episodes of frequent hypercapnic exacerbations (at least 2 over the last 12 months)

In case of restrictive diseases :

Daytime hypercapnia (PaCO2>6 kPa (kilopascal) or 45 mm Hg) or Nocturnal desaturation (SaO2 < 88%) for at least 5 minutes without obstructive sleep apnea syndrome (OSAS) found or Marker of progression of neuromuscular damage (Maximum inspiratory pressure < 60 cm H2O and forced vital capacity (FVC) less than 50% of theory)

* NIV's start from at least 6 months.
* Patient who did not object to being included in the study.
* Patient in stable condition without exacerbation (for at least 3 months)

Exclusion Criteria :

* Minor patient
* Pregnant or breastfeeding women
* Adult patient subject to enhanced protection, deprived of liberty by judicial or administrative decision.
* Patient who is physically or psychologically unable to follow the protocol in an informed manner.
* Patient with chronic respiratory failure requiring mechanical ventilation by tracheotomy
* Patient having changed center or service provider (data not available).
* Patient who objected to being included in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with chronic respiratory insufficiency fitted with long-term NIV, whatever the reason for the chronic respiratory insufficiency.
  A transcutaneous capnography within 15 days preceding the follow-up consultation and obtaining the SIM card containing the machine data will be required to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Ventilation's efficiency/tolerance | Up to 14 days
  Presence of a significant rate of patient-ventilator asynchrony when reading the ventilation curves of the NIV machine data.

SECONDARY OUTCOMES:
Estimation of quality of life with non-invasive ventilation | Up to 14 days
  Estimation of perceived quality of life through the S3-Non Invasive Ventilation questionnaire (scale from 0 to 4 ; 0 being the worst outcome)
Estimation of quality of sleep with non-invasive ventilation | Up to 14 days
  Estimation of perceived quality of sleep through the Epworth sleepiness scale (scale from 0 to 3 ; 3 being the worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: JAFFRE, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided